CLINICAL TRIAL: NCT02318615
Title: The Efficacy and Safety of Immediate Axillary Plasty With Pedicled Partial Latissimus Dorsi Muscle Flap for Lymphedema Prevention in Breast Cancer Patients Who Undergoing Axillary Dissection: a Prospective, Corhort Study
Brief Title: Immediate Axillary Plasty With a Pedicled Muscle Flap for Breast Cancer Related Lymphedema Prevention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AxLD; PKUPHBR001 (Other: PKUPH)
Record Dates: First submitted 2014-12-11; First posted 2014-12-17 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Lymphedema; Breast Neoplasm
Keywords: Breast Neoplasm; Lymphedema; Autologous flap; lattismus dorsi flap
MeSH Terms: conditions — Lymphedema; Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Axillary Plasty (Experimental): Immediate Axillary Plasty ：After axillary lymph node dissection, a pedicled flap named Partial Latissimus Dorsi Muscle Flap is filled in the cavity of axilla, and fixed around the axillary vessels.
  Interventions: Procedure: Immediate Axillary Plasty
- Education (No Intervention): Education：After surgery, education on the prevention of lymphedema. In patients suffering with upper limb lymphedema during follow-up, any treatment except axillary or breast reconstruction can be used.

INTERVENTIONS:
Procedure: Immediate Axillary Plasty — Immediate Axillary Plasty would be performed to reduce the formation of scar in the axilla.
  Arms: Immediate Axillary Plasty

SUMMARY:
The purpose of this comparable cohort study is to evaluate the efficacy and safety of immediate axillary plasty with pedicled partial Latissimus Dorsi muscle flap for lymphedema prevention in breast cancer patients who are undergoing axillary dissection.

DETAILED DESCRIPTION:
Upper limb lymphedema is the main complication of axillary dissection. It is estimated that as many as 50% of patients undergoing lymph node dissection go on to develop lymphedema, with significantly decreased quality of life with frequent infections, decreased range of motion, and a cosmetic deformity. The treatment of lymphedema was be frustrated by technical difficulties and gave rise to a heavy budget burden. Some retrospective studies revealed that immediate and delayed breast reconstruction with lattismus dorsi flap brought unexpected relief to the upper limb lymphedema. The current study was composed to assess whether transferring a pedicled partial latissimus dorsi muscle flap to the axilla would prevent the occurrence of post-mastectomy lymphedema.

This prospectively designed cohort study have two parallel arms. Patients undergoing axillary dissection would be recruited to one of the two groups, according their own preference.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing axillary lymph node dissection

Exclusion Criteria:

* Prior iplateral upper limb edema
* Plan for breast or axillary reconstruction
* The thoracodorsal vessel damage
* Muscle flap volume too low

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of lymphedema and/or severity of lymphedema | Up to 3 years

SECONDARY OUTCOMES:
Shoulder Mobility | up to 3 years
  Shoulder Mobility： the difference between baseline and postoperation，including flexion extension rotation abduction and adduction.
Postoperation seroma | up to one month
  The incidence of axilla and donor site
Acute Upper limb thrombosis | Up to one month
  The incidence of thrombosis linked to postoperation immobility

CONTACTS AND LOCATIONS:
Overall Officials: Houpu Yang, MD, Principal Investigator — Peking University People's Hospital